CLINICAL TRIAL: NCT06495476
Title: Study on Ginkgo Biolba Extract Fifty in the Treatment of Mild Cognitive Impairment Associated With Cerebral Small Vessel Disease
Brief Title: Study on Ginkgo Biolba Extract Fifty and Mild Cognitive Impairment Associated With CSVD
Acronym: GRACE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2024-090-01
Record Dates: First submitted 2024-06-16; First posted 2024-07-10 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This trial was a randomized, multicenter, double-blind, placebo-controlled parallel trial. Participants were randomly assigned according to the ratio of the experimental group: control group =1:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial is a double-blind design using simulants to ensure blinding. In order to ensure the unbiased clinical operation, observation, and evaluation of this trial, a centralized randomization system will be used to achieve the allocation of subject random numbers and therapeutic drugs.
  The simulants are consistent with the corresponding subject medications in terms of specifications, appearance, packaging, labeling, and marking, and are labeled for clinical trial use.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginkgo biloba extract 50 dropping pills treatment group (Active Comparator): Ginkgo biloba extract 50 dropping pills, oral administration, 8 dropping pills /time, 3 times/day
  Interventions: Drug: Ginkgo biloba extract 50 dropping pills
- Ginkgo biloba extract 50 dropping pills Simulant treatment group (Placebo Comparator): Ginkgo biloba extract 50 dropping pills simulant, oral administration, 8 dropping pills /time, 3 times/day
  Interventions: Drug: Ginkgo biloba extract Ginkgo biloba extract 50 Drops simulant

INTERVENTIONS:
Drug: Ginkgo biloba extract 50 dropping pills — Composition: Ginkgo ketone ester, excipient polyethylene glycol 6000. Size: 10mg ginkgolides/pill.
  Arms: Ginkgo biloba extract 50 dropping pills treatment group
Drug: Ginkgo biloba extract Ginkgo biloba extract 50 Drops simulant — Composition: The main ingredient is polyethylene glycol 6000 + caramel pigment, placebo and ginkgolide drops are basically the same in color, odor and appearance.
  Size: 10 mg analog ingredient/pill.
  Arms: Ginkgo biloba extract 50 dropping pills Simulant treatment group

SUMMARY:
This study aimed to explore the efficacy and safety of Ginkgo Biolba Extract fifty in treating mild cognitive impairment associated with cerebral small vessel disease (CSVD). Subjects included based on eligibility criteria were randomized into treatment and control groups. Patients will receive the drug or placebo for 12 months. Patients were followed at baseline and at 3 months, 6 months, and 12 months after randomization. The primary outcome was the difference from baseline in the Montreal Cognitive Assessmen (MoCA) score at 12 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-75 years old, with no limitation on sex.
2. Head MRI showed SVD lesions. High white matter signal, Fazekas score ≥2 and meet one of the following requirements:

   Have ≥2 vascular risk factors (hypertension, hyperlipidemia, diabetes, current smoking); Combined lacunar foci; Combined with a new subcortical lacunar infarction (within 7 days of onset);
3. Mild vascular cognitive impairment (memory and/or other cognitive domain abnormalities lasting for at least 3 months) with a score of 18 ≤MoCA score < 26.
4. Insufficient cognitive impairment to affect independence of life (mRS≤2).
5. After enrollment, you can live in the local stable for more than two years.
6. Sign the informed consent form.

Exclusion Criteria:

1. Known or suspected allergy to the components of the investigational drug or allergic constitution.
2. With other brain diseases: Alzheimer's disease, Lewy body dementia, Parkinson's disease frontotemporal dementia, Crohn's disease, as well as other diseases that can lead to cognitive impairment, such as subdural hematoma, communicating hydrocephalus, brain tumors, drug poisoning, alcoholism, thyroid disease, and vitamin deficiency.
3. Previous diagnosis of genetic/degenerative/inflammatory related small cerebral vascular diseases, such as CADASIL, CARASIL, etc.
4. Concomitant with major depressive disorder (≥24 score in HAMD-17) or other transient organic psychosis (e.g., schizophrenia) that meets DSM-V criteria.
5. Any medication used to treat cognitive impairment in the 4 weeks prior to randomization.
6. Combined with severe neurological impairment, such as convenient hand hemiplegia, aphasia, auditory and visual impairment, the relevant examination or scale evaluation can not be completed.
7. Combined with severe gastrointestinal diseases such as indigestion, gastrointestinal obstruction, gastric and duodenal ulcers that can affect drug absorption, or inability to swallow medication.
8. Liver enzymes (ALT, AST)>2 times the upper limit of normal value, creatinine>1.2 times the upper limit of normal value, and decreased glomerular filtration rate (<90ml/min).
9. Life expectancy < 1 year, or other reasons for not being able to complete follow-up.
10. Pregnant or lactating women, or those with fertility plans.
11. Has participated in other clinical trials.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montreal Cognitive Assessment Scale | At 12months±14days after randomization.
  Montreal Cognitive Assessment Scale (Beijing Edition) scores from 0 to 30. A higher score indicates better cognitive function.

SECONDARY OUTCOMES:
Change from baseline in Montreal Cognitive Assessment Scale | At 3months±7days and 6months±14days after randomization.
  Montreal Cognitive Assessment Scale (Beijing Edition) scores from 0 to 30. Higher score indicates better cognitive function.
Changes from baseline in total cerebral small vessel disease burden | At 12months±14days after randomization.
  The severity of periventricular WMH (PV-WMH) and the deep-WMH were rated by Fazekas rating scale. The numbers of lacune and cerebral microbleed (CMB) will be collected. Perivascular spaces (PVS) in the basal ganglia was rated with the semi-quantitative rating scale developed by the Edinburg group. Total CSVD burden was the sum of points awarded for the presence or absence of four MRI markers: one point was awarded if lacunes were present, one point was awarded if CMBs were present, one point was awarded if there were moderate to severe PVS (>10) in the basal ganglia, and one point was awarded for either confluent deep WMH (Fazekas scale 2 or 3) or irregular PV-WMH extending into the deep white matter (Fazekas score 3).
Changes from baseline in Mini-mental State Examination score | At 3months±7days, 6months±14days and 12months±14days after randomization.
  Mini-mental State Examination (MMSE) scores from 0 to 30. A higher score indicates better cognitive function.
Change from baseline in the Ability Daily Living score | At 3months±7days, 6months±14days and 12months±14days after randomization.
  Ability Daily Living (ADL) scores from 14 to 56. A higher score indicates a worse ability of daily living.
Change from baseline in Social functioning questionnaire | At 3months±7days, 6months±14days and 12months±14days after randomization.
  Social functioning questionnaire (FAQ) scores from 0 to 30. A higher score indicates a worse capacity of action.
Change from baseline in biomarkers | At 3months±7days, 6months±14days and 12months±14days after randomization.
  Biomarkers including hs-CRP, IL-6, TNF-α, Hcy, D-dimer, Fib